CLINICAL TRIAL: NCT05200780
Title: Standardization of Quantitative Muscle Ultrasonographic Parameters Among Egyptian Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Soliman Abd elhafeez, Standardization of quantitative muscle ultrasonographic parameters among Egyptian population, Assiut University
Other Study IDs: muscle ultrasonography
Record Dates: First submitted 2022-01-01; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Muscle Disease
MeSH Terms: conditions — Muscular Diseases | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasound — All subjects will undergo the tests with the same machine. Transverse ultrasound images were obtained using the Philips HD with a 4-12 MHz probe. in neurosonology unit in neurology department.

SUMMARY:
1-standardization of semi quantitative muscle ultrasonographic parameters ( muscle thickness (MT) and echo intensity (EI) ) in healthy adults and to obtain a set of normal values of all accessible muscle in both upper and lower limbs.

2.standardizaition of quantitative muscle ultrasonographic parameters (Gray scale level (GSL), Calibrated muscle backscatter values (cMBs), Optical Density (OD), 2D Textu1) in healthy adults and to obtain a set of normal values of all accessible muscle in both upper and lower limbs.

DETAILED DESCRIPTION:
. Ultrasound is a widely used imaging technique in many different medical specialties. It is a non-invasive, safe and relatively cheap investigation method.

Ultrasound is a non-invasive method to quantitatively measure various muscle parameters.

Ultrasound imaging (US) has shown to be capable of visualizing normal and pathological skeletal muscles.(1) By measuring muscle thickness (MT) and echo intensity (EI) (=grey-value) of the muscle, structural changes caused by neuromuscular disorders can be detected. (2, 3, 4) Quantitative evaluation of US images is preferable over visual evaluation, because it is more sensitive and objective and offers the possibility to perform statistical analysis.(5) A prerequisite for the diagnostic use of quantitative muscle US is the availability of normal reference values.

Ultrasonography can detect structural muscle changes caused by neuromuscular disease. Quantitative analysis is the preferred method to determine if ultrasound findings are within normal limits, but normative data are incomplete.(6)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects were recruited amongst colleagues and family members of the researchers
2. Age group (5-70)years
3. Male and female.

Exclusion Criteria:

1. Patient refuse to participate
2. The anatomy is altered due to sever trauma,tumor,or surgery

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Healthy subjects were recruited amongst colleagues and family members of the researchers
  2. Age group (5-70)years
  3. Male and female.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
get a refrence for ultrasonographic parameters muscle | 10 months
  1. use new, easy ,non-invasive tool "neuromuscular ultrasound"
  2. ultrasound give important morphological information of the muscles and can differentiate normal and diseased muscle.
  1_use new, easy ,non-invasive tool "neuromuscular ultrasound" 2_ultrasound give important morphological information of the muscles and can differentiate normal and diseased muscle.1_use new, easy ,non-invasive tool "neuromuscular ultrasound" 2_ultrasound give important morphological information of the muscles and can differentiate normal and diseased muscle.

SECONDARY OUTCOMES:
detect early pathological changes in muscles | 8 months
  Ultrasonography give pathophysiological insights and substantially added to diagnostic accuracy and treatment decisions amongst myopathies

CONTACTS AND LOCATIONS:
Overall Officials: Ghaydaa Ahmed shehata, prof, Principal Investigator — medical service affiliation

REFERENCES:
- [Background] Heckmatt JZ, Dubowitz V, Leeman S. Detection of pathological change in dystrophic muscle with B-scan ultrasound imaging. Lancet. 1980 Jun 28;1(8183):1389-90. doi: 10.1016/s0140-6736(80)92656-2. PMID 6104175
- [Background] Reimers CD, Schlotter B, Eicke BM, Witt TN. Calf enlargement in neuromuscular diseases: a quantitative ultrasound study in 350 patients and review of the literature. J Neurol Sci. 1996 Nov;143(1-2):46-56. doi: 10.1016/s0022-510x(96)00037-8. PMID 8981297
- [Background] Pillen S, Verrips A, van Alfen N, Arts IM, Sie LT, Zwarts MJ. Quantitative skeletal muscle ultrasound: diagnostic value in childhood neuromuscular disease. Neuromuscul Disord. 2007 Jul;17(7):509-16. doi: 10.1016/j.nmd.2007.03.008. Epub 2007 May 29. PMID 17537635
- [Background] Walker FO, Cartwright MS, Wiesler ER, Caress J. Ultrasound of nerve and muscle. Clin Neurophysiol. 2004 Mar;115(3):495-507. doi: 10.1016/j.clinph.2003.10.022. PMID 15036045
- [Background] Pillen S, van Keimpema M, Nievelstein RA, Verrips A, van Kruijsbergen-Raijmann W, Zwarts MJ. Skeletal muscle ultrasonography: Visual versus quantitative evaluation. Ultrasound Med Biol. 2006 Sep;32(9):1315-21. doi: 10.1016/j.ultrasmedbio.2006.05.028. PMID 16965971
- [Background] Arts IM, Pillen S, Schelhaas HJ, Overeem S, Zwarts MJ. Normal values for quantitative muscle ultrasonography in adults. Muscle Nerve. 2010 Jan;41(1):32-41. doi: 10.1002/mus.21458. PMID 19722256